CLINICAL TRIAL: NCT01145781
Title: Randomised Intervention Trial to Evaluate Single- and Double- Freeze Cryotherapy in the Prevention of Cervical Neoplasia
Brief Title: Trial to Evaluate Single- and Double- Freeze Cryotherapy in the Prevention of Cervical Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Gauravi Ashish Mishra, Associate professor Department of Preventive Oncology, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 649
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: ectocervical CIN lesions
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-freeze cryotherapy (Active Comparator): Arm 1 Single-freeze technique; 3 minutes of freeze and 5 minutes of thaw.
  Interventions: Procedure: Cryotherapy
- Double-freeze cryotherapy (Active Comparator): Arm 2 Double-freeze technique: 3 minutes of freeze and 5 minutes of thaw and cycle repeated once again.
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Cryotherapy — Arm 1 Single-freeze technique; 3 minutes of freeze and 5 minutes of thaw. Arm 2 Double-freeze technique: 3 minutes of freeze and 5 minutes of thaw and cycle repeated once again.

SUMMARY:
To evaluate whether single- and double-freeze cryotherapy techniques have similar efficacy in controlling different grades of cervical intraepithelial neoplasia (CIN), and have similar side effects and complications.

DETAILED DESCRIPTION:
Healthy women aged 25 to 64 yrs with histology confirmed ectocervical CIN lesions confined to ectocervix without extension to endocervix or vagina will be randomized to single- or double-freeze cryotherapy, as per the inclusion criteria will be invited to participate in the study.

They will be explained about the study. Informed consent will be obtained from each recruited woman. The cases selected with lesions that can be adequately covered with largest cryo probe (2.5 cm diameter) will be randomized between the following arms.

Arm 1 Single-freeze technique; 3 minutes of freeze and 5 minutes of thaw. Arm 2 Double-freeze technique: 3 minutes of freeze and 5 minutes of thaw and cycle repeated once again.

The patients will be advised about excessive discharge per vagina for 4 weeks and mild abdominal cramps.

They will be advised to abstain from sexual intercourse for 6 weeks. They would be followed up after one month for clinical evaluation and at 12th month to determine the cure rates by Pap test, HPV Test and colposcopy with or without biopsy.

The reference investigations to determine cure rates at the end of 12 months would be Pap smear, HPV Testing by HC II and colposcopy with or with out biopsy which will be offered to all the participants and biopsy will be done on women with colposcopic abnormalities.

Randomized trial: Stratified by lesion. Randomisation and analysis will be stratified on the grades of CIN.

Randomisation process:

Each woman eligible for cryotherapy who presents for treatment, will be allocated a randomisation number.

This randomisation number is a 4 digit number: The first digit represent the CIN stage (1, 2 or 3), the 3 next digits are the sequential number of the patient (from 001 to 999). Each sequential number is randomly attributed to a treatment arm. The table containing this information will be kept by the principal investigator and is only known by the people involved in the treatment.

The arm the patient has been randomised to will not be known by the people performing the follow-up visit in order to avoid any reporting bias. As soon as the patient has been randomised to double- or single-freeze, the box corresponding to the sequential number line and the CIN column will be marked with 'X'. The randomisation protocol will be rigorously followed.

Women with biopsy proven ASCUS-H and CIN lesion, after obtaining an informed consent will be randomized between single and double freeze treatment cases. The first follow-up is after one month and the next at 12th month, where patient would be subjected to Pap test, HPV Test by Hybrid Capture II and colposcopy with or without biopsy.

ELIGIBILITY:
Inclusion Criteria Apparently healthy women aged 25 to 64 yrs with following criteria will be eligible to participate in the study.

1. Histological confirmation of ASCUS -H, CIN I, CIN II and CIN III lesions.
2. The lesion confined to ecto cervix only.
3. No obvious cervical and vaginal infection.
4. Women in proliferative phase of menstrual cycle or post menopausal cases.
5. Negative endo cervical curettage.

Exclusion criteria Women less than 25 and more than 64 years will not be enrolled.

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary end point is the cure rate at the end of one year | 1 year
  The primary end point is the cure rate at the end of one year by comparing between two different techniques of cryotherapy i.e. single freeze and double freeze.

SECONDARY OUTCOMES:
The secondary end points are the rates and the types of side effects and complications | 1 year
  The secondary end points are the rates and the types of side effects and complications by comparing between two different techniques of cryotherapy i.e. single freeze and double freeze.

CONTACTS AND LOCATIONS:
Overall Officials: Gauravi A MIshra, MD, Principal Investigator — Tata Memorial Hospital; Sharmila A Pimple, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided